CLINICAL TRIAL: NCT06682078
Title: DEV-GEN-RiTuGo - Assessment of Individual Gonadal Tumor Risk in Patients With Disorders of Sexual Developpment According to the Etiology.
Brief Title: Disorders of Sexual Development and Gonadal Tumor Risk
Acronym: DEV-GEN-RiTuGo
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0858; 23-5235 (Registry Identifier: GDPR)
Record Dates: First submitted 2023-08-22; First posted 2024-11-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: Disorders of Sexual Development
Keywords: surgery; pediatrics; Urology; Endocrinology; Gonadoblastoma; Dysgerminoma; neoplasms; gonadal tissue; sexual development; oncology; gonadal dysgenesis; androgen-insensitivity syndrome; testicular regression syndrome; anti-mullerian hormone
MeSH Terms: conditions — Disorders of Sex Development; Gonadoblastoma; Dysgerminoma; Neoplasms; Gonadal Dysgenesis; Androgen-Insensitivity Syndrome; Anorchia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Not applicable . Non-interventional retrospective study, only on datas. — Not applicable . Non-interventional retrospective study, only on datas.

SUMMARY:
Disorders of Sexual Development are rare and represent a spectrum of heterogeneous pathologies. The risk of developing a malignant gonadal germ cell tumor (MGCT) exists and varies according to the etiology.

The indication for prophylactic gonadectomy must be modulated and discussed for all patients. It is essential to assess each patient's individual risk.

The aim of our study is to assess gonadal tumor risk in patients with Disorders of Sexual Development according to etiology

The primary objective is to evaluate tumor risk and the indication for gonadectomy in cases of Disorders of Sexual Development according to etiology.

The secondary objectives are to evaluate the timing of gonadectomy, to monitor changes in practice over time, and to assess the contribution of imaging and/or biological tests to tumor detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent gonadectomy for variation in genital development between 1990 and 2022.
* Pathological anatomy examination in Lyon
* With clinical data
* With karyotype
* 3 categories:

  * with genetic diagnosis
  * without genetic diagnosis because searched but not found
  * without genetic diagnosis because not searched

Exclusion Criteria:

* Biopsies without gonadectomy
* Fetus
* Operated outside the period 1990-2022
* Lack of clinical data
* No karyotype

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients who underwent gonadectomy for Disorders of Sexual Development between 1990 and 2022, followed by Dr. Daniela Gorduza in the Pediatric Uro-Visceral Surgery Department of the hospital Femme-Mère-Enfant.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of gonadal tumor lesion after gonadectomy, in case of Disorders of sexual development (DSD) according to anatomo-pathological analysis. | The outcome measure will be assessed and the datas reported for each patient will be collected, from birth until the study completion date, or by default until the date of death from any cause. Datas will be collected during the 10 months of the study
  Datas about the gonadectomy surgical pieces performed between1990 and 2022 are reviewed for the study by Dr Frédérique Dijoud, anatomo-pathologist at the DEV-GEN CRMR in Lyon, to confirm the présence or absence of a gonadal tumor lesion, in order to avoid intra- and inter-reader interpretation bias.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie uro-viscérale pédiatrique, Bron, France

IPD SHARING:
Plan to Share IPD: No